CLINICAL TRIAL: NCT02397499
Title: A Multi-Center, Randomized, Double-Blinded, Placebo-Controlled Study Evaluating the Safety and Efficacy of LIPO-202 for the Reduction of Central Abdominal Bulging Due to Subcutaneous Fat in Non-Obese Subjects
Brief Title: Evaluating the Safety and Efficacy of LIPO-202 for the Reduction of Central Abdominal Bulging Due to Subcutaneous Fat
Acronym: AbCONTOUR1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Neothetics, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LIPO-202-CL-18
Record Dates: First submitted 2015-03-19; First posted 2015-03-25 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Central Abdominal Bulging
MeSH Terms: interventions — Salmeterol Xinafoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- LIPO-202 (Experimental): Experimental arm
  Interventions: Drug: LIPO-202
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: LIPO-202
  Other Names: Salmeterol
  Arms: LIPO-202
Drug: Placebo
  Other Names: Placebo for LIPO-202
  Arms: Placebo

SUMMARY:
This is a multi-center, randomized, double-blinded, placebo-controlled study evaluating the safety and efficacy of LIPO-202 for the reduction of central abdominal bulging due to subcutaneous fat in non-obese subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or non-pregnant female subjects
* Capable of providing written consent.
* BMI < 30 kg/m2
* Stable diet and exercise routine
* Central abdominal bulging that is evaluated by the clinician at least slight bulge, not flat

Exclusion Criteria:

* Have had any treatment of the fat around your abdomen, including surgical procedures (tummy tuck, liposuction), injections for fat loss or treatments with devices to reduce fat in your abdomen.
* Plan on starting a weight loss or exercise program during the study.
* Known hypersensitivity to study drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 800 (Estimated)
Dates: Start 2015-04; Primary Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Safety as measured by Physical examination, adverse events, vital signs, and laboratory tests. | 8 weeks
  Physical examination, adverse events, vital signs, and laboratory tests.
Change in the clinician reported photonumeric score | 8 weeks post the start of treatment
Change in the patient reported global abdominal perception score | 8 weeks post the start of treatment

SECONDARY OUTCOMES:
Change in waist circumference | 8 weeks post the start of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Maria Feldman, Study Director — Neothetics, Inc
Locations (31):
- United States (31):
  - WG Clinical Research, Tucson, Arizona
  - Burke Pharmaceutical Research, Hot Springs, Arkansas
  - Clinical Testing Center of Beverly Hills, Beverly Hills, California
  - Center for Dermatology Cosmetic and Laser Surgery, Fremont, California
  - Dermatology/Cosmetic Laser Associates of La Jolla, Inc, San Diego, California
  - University Clinical Trials, Inc., San Diego, California
  - Clinical Science Institute, Santa Monica, California
  - The Center for Clinical & Cosmetic Research, Aventura, Florida
  - Skin Care Research, Inc., Boca Raton, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - International Dermatology Research, Miami, Florida
  - Altman Dermatology Associates, Arlington Heights, Illinois
  - Glazer Dermatology, Buffalo Grove, Illinois
  - Dermatology Specialists Research, Louisville, Kentucky
  - Grekin Skin Institute, Warren, Michigan
  - Minnesota Clinical Study Center, Fridley, Minnesota
  - Skin Specialists, PC, Omaha, Nebraska
  - Skin Laser & Surgery Specialist of NY/NJ, Hackensack, New Jersey
  - Juva Skin & Laser Center, New York, New York
  - Skin Specialty Dermatology, New York, New York
  - Marina I Peredo, M.D, P.C., Smithtown, New York
  - Aesthetic Solutions, Chapel Hill, North Carolina
  - Dermatology, Laser and Vein Specialists of the Carolinas, Charlotte, North Carolina
  - Westlake Dermatology Clinical Research Center, Austin, Texas
  - J & S Studies, Inc., College Station, Texas
  - Menter Dermatology Research Center, Dallas, Texas
  - Suzanne Bruce and Associates, P.A., The Center for Skin Research, Katy, Texas
  - Research Across America, Plano, Texas
  - Dermatology Research Center, Inc., Salt Lake City, Utah
  - Virginia Clinical Research, Inc., Norfolk, Virginia